CLINICAL TRIAL: NCT00427765
Title: A Phase II Study of High-Dose Intravenous Busulfan Plus Melphalan With Allogeneic or Autologous Marrow or Peripheral Blood Progenitor Cell Transplantation for Lymphoid Malignancies or Multiple Myeloma
Brief Title: Busulfan Plus Melphalan Conditioning Regimen for Lymphoid Malignancies or Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0190
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-12

CONDITIONS: Multiple Myeloma; Lymphoma
Keywords: Multiple Myeloma; Hodgkin's Disease; Non-Hodgkin's Lymphoma; Leukemia; Lymphoma; Busulfan; Melphalan; Autologous bone marrow; BMT; Peripheral blood stem cell transplant; PBSCT
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia | interventions — Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan + Melphalan (Experimental): Busulfan 32 mg/m^2 intravenous (IV) for 1 Day then 130 mg/m^2 IV for 4 Days; and Melphalan 70 mg/m^2 IV for 2 Days
  Interventions: Drug: Busulfan; Drug: Melphalan

INTERVENTIONS:
Drug: Busulfan — Test Dose = 32 mg/m^2 IV for 1 Day; 130 mg/m^2 IV for 4 Days
  Other Names: Busulfex
Drug: Melphalan — 70 mg/m^2 IV for 2 Days

SUMMARY:
Primary Objectives:

1. To determine the efficacy of administering multiple doses of intravenous (i.v.) busulfan at a dose of 130 mg/m2, to yield a systemic plasma drug exposure represented by a daily area under the plasma concentration versus time curve (AUC) of approximately 5,000 mMol-min for 4 days, followed by i.v. melphalan at a dose of 70 mg/m2 for 2 days in adult patients receiving autologous or allogeneic transplantation for lymphoid malignancies or myeloma.
2. To describe the plasma pharmacokinetic (PK) profiles of busulfan and melphalan in this regimen.
3. To determine the disease-free and overall survival of patients receiving this preparative regimen.
4. To determine the treatment-related morbidity and mortality of this combination of drugs.

DETAILED DESCRIPTION:
Busulfan and melphalan are both traditional alkylating agents that are designed to interfere with the production of cancer cells at the DNA (deoxyribonucleic acid) and RNA (ribonucleic acid) level.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete physical exam, including routine blood (2-3 teaspoons) and urine tests. Patients will have a chest x-ray, heart scan, lung function test, and a bone marrow biopsy. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will be able to start receiving chemotherapy treatment with busulfan and melphalan. Participants who agree to the optional blood draws described above will at first receive a therapeutic "trial dose" of busulfan by vein to test the blood levels over time. This therapeutic trial dose of busulfan is about 25% (1 fourth) of the full therapeutic dose of the drug. This information will be used to decide what the future high-dose busulfan treatments you receive will be. If you do not agree to the optional blood draw, you will receive a fixed amount of high-dose busulfan from the start.

On the 1st day of hospitalization, you will receive fluids by vein through a central venous catheter. If you choose the optional busulfan dose for pharmacokinetic-based busulfan dosing, you will receive the optional busulfan dose 9 days before stem cell infusion (Day 1), followed by a rest day on Day 2. If you choose to receive a fixed dose of busulfan, busulfan will be injected through a central venous catheter over 3 hours, once a day, for the next 4 days (Days 3-6, ending 3 days before the stem cell infusion day).

Patients receiving pharmacokinetic-based dosing of busulfan will also continue to receive busulfan on Days 3-6. This will be followed by melphalan for all patients, given through your central venous catheter over 30 minutes, once a day, for 2 days, on days 8 and 9. Your stem cell infusion day will be on Day 10 of treatment.

Patients receiving 5 out of 6 antigen matched-related allogeneic stem cell transplants or unrelated allogeneic stem cell transplants will also receive antithymocyte globulin (ATG), by vein, on Days 7-9, up to one day before the stem cell infusion. This is given to decrease the risk of GVHD and graft rejection in mismatched transplants.

On Day 10, healthy blood stem cells or bone marrow from the donor will be given through the central catheter. This is your transplant date. You will also receive several other medications to help the treatment work and to help prevent infections while your immune system is weak. Tacrolimus and methotrexate will be given to decrease the risk of graft-versus-host-disease (GVHD). GVHD occurs when the donor's immune cells fight the patient's body. The tacrolimus will be started on the day before the transplant and will continue for up to six months. Tacrolimus is given by vein at first and then by mouth when you are able to eat. Methotrexate is given by vein on Days 11, 13, 16, and possibly on Day 21, up to 11 days after the transplant.

Please note that the treatment dates listed above were used to help explain your general treatment plan. By standard medical convention, the day of stem cell infusion is always listed as day zero. Therefore, the days listed above are different from the treatment plan described in the protocol and abstract.

Sulfamethoxazole (Bactrim) or pentamidine will be given to fight bacteria. Bactrim is given by mouth when the counts are good. Pentamidine is given by vein when the counts are low. Acyclovir will be given at first by vein and then Valtrex (valacyclovir) will be given by pill to decrease the risk of viral infections. Granulocyte colony-stimulating factor (G-CSF) will be given to help the new bone marrow grow. It is given as an injection under the skin after the transplant. It will continue until the white blood cells reach an acceptable level. Overall, some of these drugs will be given for as long as 6 months or possibly longer. Other medications may be necessary. If you are allergic to some of these drugs, changes will be made.

You will be in the hospital for about 3-4 weeks. You will have checkups every day until discharged from the hospital. You will then be seen in the outpatient clinic at least 3 times a week until your blood counts improve. You will be seen by your doctor at least every week until 100 days after the bone marrow transplant. You must stay in Houston during this time. After 100 days, you will return to the clinic according to your individual physician's recommendations.

Some patients may need to receive spinal taps with instillation of chemotherapy several times over the year after transplantation. This is only for patients with a previous clinical history of leukemic involvement of the brain or high risk of developing leukemia relapse in the brain. The spinal tap is performed in the clinic. You are given local anesthetic at the lower back site, a small needle is inserted in the space between 2 spinal bones, a small amount of fluid that bathes the brain (cerebrospinal fluid) is removed for testing, and a small amount of chemotherapy is given.

Bone marrow samples will be taken at about 1 month and 3 months after the transplant. You will also have a lung function test at 3 months after the transplant.

This is an investigational study. The FDA has approved all of the drugs used in this study for use in stem cell transplantation. Up to 168 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoid malignancies, including Hodgkin's and non-Hodgkin's lymphoma (primary refractory or recurrent), or multiple myeloma (beyond first complete remission or unresponsive to therapy. Complete remission for multiple myeloma defined by absence of detectable paraprotein in serum and/or urine by immunoelectrophoresis or immunofixation, and < 5% plasma cells in the bone marrow), not qualifying for treatment protocols of higher priority.
* Age 18 to 65 years of age.
* Adequate renal function as defined by estimated serum creatinine clearance > 50 ml/min and serum creatinine < 1.8 mg/dL.
* Adequate hepatic function, as defined by serum glutamic pyruvic transaminase (SGPT) < 3 * upper limit of normal; serum bilirubin and alkaline phosphatase < 2 * upper limit of normal, or considered not clinically significant.
* Adequate pulmonary function with Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and Capacity of the Lung for Carbon Monoxide (DLCO)> 50%. Exceptions may be allowed for patients with pulmonary involvement after discussing with principal investigator (PI).
* Adequate cardiac function with left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
* Zubrod performance score < 2.
* Patients receiving an allogeneic transplant must have an HLA matched, or one A, B, or DR mismatched related donor. Unrelated donor must be matched at A, B, and DR (defined as A, B serologic matched and DRB1 molecular matched). Donor must be willing to donate peripheral blood or bone marrow progenitor cells.
* Patient and donor should be willing to participate in the study by providing written consent.
* Female patient must not be pregnant and have negative pregnancy.

Exclusion Criteria:

* Patients with unresolved grade >/= 3 non-hematologic toxicity from previous therapy. Patients with grade 2 toxicity will be eligible at the discretion of the PI.
* Patients with active Central Nervous System (CNS) disease.
* Evidence of acute or chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Study Chairman and consider liver biopsy.
* Uncontrolled infection, including Human immunodeficiency virus (HIV) or Human T-lymphotropic virus Type I (HTLV-1) infection.
* Patients who have had a previous autologous or allogeneic stem cell transplant during the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2004-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nieto Y, Gruschkus S, Valdez BC, Jones RB, Anderlini P, Hosing C, Popat U, Qazilbash M, Kebriaei P, Alousi A, Saini N, Srour S, Rezvani K, Ramdial J, Barnett M, Gulbis A, Shigle TL, Ahmed S, Iyer S, Lee H, Nair R, Parmar S, Steiner R, Dabaja B, Pinnix C, Gunther J, Cuglievan B, Mahadeo K, Khazal S, Chuang H, Champlin R, Shpall EJ, Andersson BS. Improved outcomes of high-risk relapsed Hodgkin lymphoma patients after high-dose chemotherapy: a 15-year analysis. Haematologica. 2022 Apr 1;107(4):899-908. doi: 10.3324/haematol.2021.278311. PMID 33951890
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2/4/2005 through 10/29/2010. All participant recruitment attempted at UT MD Anderson Cancer Center.
Pre-assignment Details: Among the participants enrolled, two were excluded from the trial before starting any treatment. There are two participants who were enrolled on the study twice (having to temporarily leave then re-enter the study).
Period: Overall Study
Arm/Group | Busulfan + Melphalan
Started | 164
Completed | 164
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan + Melphalan
Number analyzed (Participants) | 164
Age Continuous [Median (Full Range); unit: years] | 42 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 97
Region of Enrollment [Number; unit: participants]
  United States | 164

OUTCOME MEASURES:

1. Primary Outcome: Average Overall Survival Time
Description: Average number of years for survival post transplant where overall survival time is measured from date of transplant to disease progression or death for any reason.
Time Frame: Baseline(transplantation) to disease progression or death for any reason, up to 6 years.
Population: Analysis by protocol
Measure: Mean (Full Range); unit: years
Arm/Group | Busulfan + Melphalan
Number analyzed (Participants) | 164
years | 3 [0.1 to 6]

ADVERSE EVENTS:
Time Frame: 5 years and 9 months
Arm/Group | Busulfan + Melphalan
Serious Adverse Events (participants affected / at risk) | 31/164
Other Adverse Events (participants affected / at risk) | 164/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Melphalan (N=164)
Acute Renal Failure (Renal and urinary disorders) | 3 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Cholecystitis (General disorders) | 1 (1)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Graft Vs Host Disease (General disorders) | 9 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (General disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection/Sepsis (Infections and infestations) | 2 (2)
Veno-Occlusive Disease (Hepatobiliary disorders) | 1 (1)
Graft Failure (General disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Portal Vein Flow (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Melphalan (N=164)
Dysrhythmia (Cardiac disorders) | 1 (1)
Edema (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 3 (3)
Thrombotic Thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 110 (110)
Mucositis (Gastrointestinal disorders) | 138 (138)
Nausea (Gastrointestinal disorders) | 156 (156)
Elevated Creatinine (Renal and urinary disorders) | 4 (4)
Hemorrhagic Cystitis (Renal and urinary disorders) | 16 (16)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 3 (3)
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 4 (4)
Elevated Bilirubin (Hepatobiliary disorders) | 11 (11)
Veno-Occlusive Disease (Hepatobiliary disorders) | 3 (3)
Infections (Infections and infestations) | 70 (70)
Neutropenic Fever (General disorders) | 72 (72)
Confusion (General disorders) | 3 (3)
Headache (General disorders) | 3 (3)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1)
Cranial Nerve Palsy (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 3 (3)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Graft Vs Host Disease (General disorders) | 48 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No